CLINICAL TRIAL: NCT01669655
Title: Plasma Profile of Exclusively Breastfed Infants
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: AK99
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Breast Fed Infants
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample; Human Milk sample
Oversight: Data Monitoring Committee: No

SUMMARY:
To characterize nutrient levels in breastfeeding infants and their mothers.

DETAILED DESCRIPTION:
The objectives of this study are (1) to characterize plasma lutein levels in breastfed infants in an Asian population where lactating mothers have diets habitually high in lutein and (2) investigate how blood lutein levels in breastfed infants vary according to lutein content of the mothers' milk in such a population.

ELIGIBILITY:
Inclusion Criteria:

* Infant is judged to be in good health.
* Infant is a singleton from a full term birth.
* Infant's birth weight was > 2490 g.
* Infant is between 6 weeks and 16 weeks (42 to 112 days).
* Infant must have been exclusively breastfed at enrollment.
* Mother's intake indicates a consumption of an average of at least three servings of fruit and/or vegetables per day.
* Mother is a non-smoker.
* Mother is in good health.
* Mother confirms her intention to continue breastfeeding.

Exclusion Criteria:

* An adverse maternal, fetal or infant medical history that is thought to have potential for effects on growth, and/or development.
* Infants who have consumed medications or herbal preparations during past 14 days prior to enrollment.
* Infants who have consumed any solid or liquid foods or juices prior to enrollment.
* Infants who have received any supplements containing carotenoids prior to enrollment.
* Mother who is consuming dietary supplements containing carotenoids.
* Participation in another study that has not been approved as a concomitant study.

Ages: 6 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Breastfeeding infants and their mothers
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Plasma carotenoids in breastfed infants | At visit 1 (enrollment)

SECONDARY OUTCOMES:
Plasma carotenoids in mothers of breastfed infants | At visit 1 (enrollment)
Dietary carotenoid intake of mothers of breastfed infants | At visit 1 (enrollment) and visit 2 (14 days)
Carotenoid levels in breastmilk | At visit 1 (enrollment) and visit 2 (14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Xianfeng Zhao, MD, PhD, Study Chair — Abbott Nutrition, R&D China
Locations (1):
- Fudan University of Shanghai, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu X, Zhao X, Berde Y, Low YL, Kuchan MJ. Milk and Plasma Lutein and Zeaxanthin Concentrations in Chinese Breast-Feeding Mother-Infant Dyads With Healthy Maternal Fruit and Vegetable Intake. J Am Coll Nutr. 2019 Feb;38(2):179-184. doi: 10.1080/07315724.2018.1490934. Epub 2018 Sep 11. PMID 30204542